CLINICAL TRIAL: NCT05741879
Title: Gamified Exercise Intervention to Improve Children's Adherence to 24-hour Movement Recommendations in a Family-Based Health Setting: "3,2,1 Move on Crossover Study".
Brief Title: Gamified Family-based Health Exercise Intervention to Improve Adherence to 24-h Movement Behaviors Recommendations in Children.
Acronym: Move On
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pública de Navarra (Other)
Collaborators: European Regional Development Fund (Other); Gobierno de Navarra Departamento de Salud (Unknown); NavarraBiomed Biomedical Research Center (Other); Centro Atención Primaria de Iturrama (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PI_2021/111
Record Dates: First submitted 2023-02-03; First posted 2023-02-23 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2023-02

CONDITIONS: Physical Inactivity; Obesity, Childhood; Sedentary Behavior
Keywords: Lack of physical fitness; Low levels of Basic Motor Skills
MeSH Terms: conditions — Sedentary Behavior; Pediatric Obesity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gamified online exercise in a family environment (Experimental): Strength training Resistance training Flexibility training Basic motor skills training Executive function training
  Interventions: Behavioral: Gamified exercise training
- Standard care Non-supervised daily routines/activities (Active Comparator): Non-supervised daily routines/activities
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Gamified exercise training — Participants will complete a 2-days-a-week online training routine with their families: Each session will include a Warm-Up/Activation phase (3 minutes: light intensity continuous training), a Training phase (10-26 minutes: 6-12 repetitions, 20-40" of work, 10-20" recovery), and a Cool Down phase (3 minutes: static and dynamic exercises). The exercises will be different each week and will increase in length and intensity accordingly. The sessions will be supervised by the participants parent(s) and/or guardian(s).
  Arms: Gamified online exercise in a family environment
Behavioral: Standard Care — This group will be allocated to standard care and therefore no gamified online exercise training will be provided. They will continue to perform their daily routine/activities including their basic motor skills classes at school and their extracurricular sports and/or cultural activities.
  Arms: Standard care Non-supervised daily routines/activities

SUMMARY:
Physical inactivity is the fourth most important risk factor for mortality worldwide and it contributes to weight gain and obesity. On the contrary, it is established that regular physical activity is a prevention and managerial factor of these non-communicable diseases. Therefore, the goal of this study is to design and evaluate the effectiveness of a 12-week physical exercise and lifestyle improvement training program carried out in a family environment, through a web platform, and with "online" supervision. This platform will improve the physical conditioning and adherence to PE in a "family environment", and to promote good development of the child through physical activities and exercises that can be done as a family at home and/or outside.

ELIGIBILITY:
Inclusion Criteria:

* Participants without any physical or mental disorders that would prevent them from completing the assessments tests or participating in the exercise intervention program
* One parent/guardian must answer the questionnaires
* Informed consent from the participants parent(s)/guardian(s)

Exclusion Criteria:

* Participants with psychiatric disorders or chronic illness that limits their participation in physical activities
* Participants who do not comply with the established procedures
* Participants who do not understand the Spanish language

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in 24-h movement behaviors (accelerometers) sedentary time. | Baseline, 12 Week, and 24 Week
  During their visit to Navarrabiomed, participants will receive a (GENEActiv, Activinsights, Kimbolton, UK) accelerometer that will objectively measure their 24-hour movement behaviors (physical activity, sedentary behaviors, and sleep). The participants will wear the accelerometer for seven consecutive days. Additionally, this accelerometer data will be supplemented with a diary to validate sleep time and (non)wear time.

SECONDARY OUTCOMES:
Changes in body composition. | Baseline, 12 Week, and 24 Week
  Body composition measured with bioelectrical impedance (fat mass and body mass).
Changes in muscle composition. | Baseline, 12 Week, and 24 Week
  Muscle composition measured with ultrasound of the thigh/quadriceps/recto femoral.
Changes in health-related physical fitness. | Baseline, 12 Week, and 24 Week
  Health-related physical fitness measured, among other tests from the PREFIT battery, with the 20-meter shuttle run test, the handgrip test and the 4x10 speed agility test.
Changes in Basic Motor Skills. | Baseline, 12 Week, and 24 Week
  Measured with the MOBAK-KG Battery with tests such as the long jump or balance over an inverted beam. MOBAK-KG sum score ranging from 0 (lowest basic motor competencies) to 16 points (highest basic motor competencies).
Changes in 24-h movement behaviors (self-reported). | Baseline, 12 Week, and 24 Week
  Self-report of physical activity levels and sedentary behaviors in youth will assessed by the Youth Activity Profile - Spain. In this questionnaire, a rating scale is used with a score from 1 to 5 in which, in the first two sections, "1" indicates low intensity and frequency of physical activity and "5" indicates high intensity and frequency of physical activity; while, in the third section, "1" indicates a low amount of sedentary behaviors and "5" an excess of them.
Changes in executive function. | Baseline, 12 Week, and 24 Week
  Measured with "Early Tools" games (Years Toolbox YET-2017).
Changes in Child Self-Regulation & Behavior. | Baseline, 12 Week, and 24 Week
  Measured with CSBQ (Child Self-Regulation & Behavior Questionnaire). Parents will be asked to think about their child's behavior during the past 6 months, and to choose whether each statement was: Not true (1), Somewhat true (2), Certainly true (3), or Can't say (4).
Changes in quality of life. | Baseline, 12 Week, and 24 Week
  Kiddy-KINDL will be used to assess the health-related quality of life in children.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Mª Alonso Martínez, Ph.D, Study Chair — Universidad Pública de Navarra
Locations (1):
- Navarrabiomed, Universidad Pública de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Legarra-Gorgonon G, Garcia-Alonso Y, Ramirez-Velez R, Alonso-Martinez L, Izquierdo M, Alonso-Martinez AM. Assessing basic motor competences, physical fitness, and executive function in 4-5-year-old children: a longitudinal study in a primary care setting. Ital J Pediatr. 2024 May 31;50(1):108. doi: 10.1186/s13052-024-01674-1. PMID 38816854
- [Derived] Alonso-Martinez AM, Legarra-Gorgonon G, Garcia-Alonso Y, Ramirez-Velez R, Alonso-Martinez L, Erice-Echegaray B, Izquierdo M. Gamified family-based health exercise intervention to improve adherence to 24-h movement behaviors recommendations in children: "3, 2, 1 Move on Study". Trials. 2023 Aug 14;24(1):531. doi: 10.1186/s13063-023-07494-8. PMID 37580788